CLINICAL TRIAL: NCT06861842
Title: Bioequivalence Study of Lithium Carbonate 300 mg Tablets. Actilitio® in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de Atencion e Investigacion Medica (Network)
Responsible Party: Principal Investigator, Humberto Reynales MD MSc PhD, Principal investigator, Centro de Atencion e Investigacion Medica
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CGIS-BIO-001-2019; Actifarma (Other: Caimed)
Record Dates: First submitted 2025-01-23; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Healthy Donors
Keywords: bioequivalence
MeSH Terms: interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Period 1 (Active Comparator): Theralite® 300 mg
  Interventions: Drug: Theralite®; Drug: Actilitio®
- Period 2 (Active Comparator): Actilitio® 300 mg
  Interventions: Drug: Theralite®; Drug: Actilitio®

INTERVENTIONS:
Drug: Theralite® — Reference
  Other Names: lithium carbonate
Drug: Actilitio® — Test
  Other Names: lithium carbonate

SUMMARY:
A bioequivalence study of lithium carbonate will be developed in 24 healthy subjects, in fasting condition

DETAILED DESCRIPTION:
A bioequivalence study of lithium carbonate will be developed in 24 healthy subjects, in fasting condition, following the design:

Open-label, crossover, randomized, single-dose design of 300 mg lithium carbonate immediate release tablets, with two treatments, two periods, two sequences in fasting condition, with a washout time of 14 days between each dose, participation as a subject in these studies implies a higher than minimal risk for the subjects.

ELIGIBILITY:
Inclusion Criteria:

* - Men or women between 18 and 50 years of age at the time of signing the informed consent form.
* Women who are unable to conceive, who are not pregnant or breastfeeding (To be considered unable to conceive, they must be at least 1 year postmenopausal or surgically sterile). Table 2.
* Female participants of childbearing capacity must be using adequate contraception for the past 6 months and agree to continue using an adequate contraceptive method for 30 days after signing the consent form
* Have been clinically diagnosed as healthy by the study physician.
* Subjects with clinical laboratory results within normal ranges and/or fit by medical screening. (Table 2)
* Subjects were non-smokers for the last 3 months at the time of screening.
* Having signed the informed consent for the study.
* Body mass index between 18-30 kg/m2.
* Subject with complete contact information (cell phone and/or landline contact, address).
* Subject who has a family member or guardian with a contact telephone number.
* Subject with the availability of time to comply with the scheduled visits and activities.
* Subject who is willing to comply with the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* - Subject diagnosed with renal, cardiac, hepatic, immunological, dermatological, endocrine, gastrointestinal, neurological, psychiatric, compulsive depressive disorder.
* Subjects with a diagnosis of hematological disorders, such as anemia and/or polycythemia.
* Subjects with history of gastric surgeries.
* Permanent or temporary use of any type of medication either on their own initiative or by medical prescription 2 days prior to the hospitalization phase of the study. Except female patients who are planning regularly with the same contraceptive method in the last 6 months prior to the beginning of the present study.
* Smoking in the last 3 months, regardless of the number of cigarettes at the time of selection.
* Drinking alcohol in excess of 16 g 15 days prior to selection as a subject, this amount being equivalent to 1 beer or 2 glasses of wine.
* Positive test for the consumption of drugs of abuse or psychoactive substances at the time of selection (Table 2).
* Known hypersensitivity to the active substance or excipients of the test product.
* Medical history of angioedema or anaphylaxis.
* Pregnant or lactating woman.
* Subject diagnosed with human immunodeficiency virus infection, hepatitis B or hepatitis C positive.
* Having participated in clinical studies in the 4 months prior to the start of the present study.
* Having donated blood or having reported blood loss greater than 500 mL in the previous 30 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
AUC | 0 hours - 72 hours
  concentration plasma under curve AUC
Cmax | 0 hours - 6 hours
  peak concentration plasma Cmax

SECONDARY OUTCOMES:
Tmax | 0 hours - 6 hours
  Pharmacokinetic Outcome Measures

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Atención e Investigación Médica, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: jul 2024 - abril 2025
Access Criteria: indicate whether a proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed
URL: https://www.caimed.com